CLINICAL TRIAL: NCT00734032
Title: A Phase II Clinical Study of SB-480848 in Dyslipidemic Patients- A Multicenter, Randomized, Double-blind, Placebo-controlled Study of SB-480848 to Evaluate the Efficacy and Safety -
Brief Title: A Phase II Clinical Study of SB-480848 in Dyslipidemic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPL110118
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Atherosclerosis
Keywords: SB-480848; Dyslipidaemia
MeSH Terms: conditions — Atherosclerosis; Dyslipidemias | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo Group (Placebo Comparator): Matched Placebo
  Interventions: Drug: SB480848 Placebo Tablet
- SB480848 40mg Group (Experimental): SB480848 40mg/day
  Interventions: Drug: SB480848 40mg EC Tablet
- SB480848 80mg Group (Experimental): SB480848 80mg/day
  Interventions: Drug: SB480848 80mg EC Tablet
- SB480848 160mg Group (Experimental): SB480848 160mg/day
  Interventions: Drug: SB480848 160mg EC Tablet

INTERVENTIONS:
Drug: SB480848 40mg EC Tablet — 1 tablet once a day
  Other Names: Darapladib
  Arms: SB480848 40mg Group
Drug: SB480848 80mg EC Tablet — 1 tablet once a day
  Arms: SB480848 80mg Group
Drug: SB480848 160mg EC Tablet — 1 tablet once a day
  Arms: SB480848 160mg Group
Drug: SB480848 Placebo Tablet — 1 tablet once a day
  Arms: Placebo Group

SUMMARY:
The primary objective of this study is to examine the effects of SB-480848 on plasma lipoprotein associated phospholipase A2 (Lp-PLA2) activity in dyslipidemic patients during a 4-week treatment with SB-480848.

ELIGIBILITY:
Inclusion criteria:

Dyslipidemic subject who is currently undergoing statin therapy and no change in lipid-lowering therapy or dose during the 4 week prior to randomization

Exclusion criteria:

1. Recent (i.e.,<6 months prior to screening) CV event and/or vascular procedure defined as:

   A)ST-elevation MI or non-ST-elevation MI B)Unstable angina C)Coronary revascularization [(percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)] D)Stroke of any etiology E)Peripheral arterial disease with critical limb ischemia (resting pain or ischemic skin lesions, either ulcers or gangrene) F)Resuscitated cardiac arrest
2. Planned CABG or planned PCI or planned major non-cardiac surgery within study period
3. No measurable Lp-PLA2 activity in plasma (<10 nmol/min/mL) at screening
4. Change in a lipid-lowering medication, regimen or dosage during the 4 week prior to randomization
5. Poorly controlled dyslipidemia (LDL-c >=160 mg/dL) at screening

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-08-26 (Actual); Primary Completion 2009-01-16 (Actual); Study Completion 2009-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL110118 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned in 100 dyslipidemic male or female participants, aged 20 to 80 years, undergoing statin therapy and no change in lipid-lowering medication or dose during the 4 weeks prior to randomization from 26 August 2008 to 16 January 2009 at 7 centers in Japan.
Pre-assignment Details: Out of 116 participants screened, 9 were screen failures; 107 participants were randomized in a ratio of 1:1:1:1, to receive placebo or any 1 of the 3 doses of SB-480848 (40 milligram [mg], 80 mg, 160 mg), prior to which they continued their statin therapy with no change in lipid-lowering medication or dose during 4 weeks of Run-in period.
Groups:
- Placebo: Participants received oral dose of matching placebo tablet once daily, after breakfast in the morning for 4 weeks of treatment period.
- SB-480848 40 mg: Participants received oral dose of SB-480848 40 mg enteric-coated tablet once daily, after breakfast in the morning for 4 weeks of treatment period.
- SB-480848 80 mg: Participants received oral dose of SB-480848 80 mg enteric-coated tablet once daily, after breakfast in the morning for 4 weeks of treatment period.
- SB-480848 160 mg: Participants received oral dose of SB-480848 160 mg enteric-coated tablet once daily, after breakfast in the morning for 4 weeks of treatment period.
Period: Overall Study
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg
Started | 25 | 28 | 28 | 26
Completed | 25 | 27 | 28 | 26
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg | Total
Number analyzed (Participants) | 25 | 28 | 28 | 26 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (11.71) | 59.8 (10.17) | 58.3 (9.54) | 58.3 (10.48) | 59.0 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 18 | 13 | 65
  Male | 8 | 11 | 10 | 13 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 25 | 28 | 28 | 26 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Plasma Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activity
Description: Blood sample for Lp-PLA2 activity was collected before administration of study medication on the sampling day. Participants were instructed to visit without meal and study medication in the morning. The study medication was administered with food following test. Baseline value was defined as the assessment done on Week 0 (Visit 2). Change from Baseline was calculated as the post-Baseline (Week 4) assessment value minus the Baseline assessment value. If either value was missing, then the change from Baseline was set to be missing. The natural logarithm (log) was used for transformation in Lp-PLA2 activity. In case of zero values, an offset of 0.0001 was added to the zero values to ensure that the log transformation was successfully applied. The log transformation was conducted on the original value and then taken the change from Baseline on that log original value, calculated as log (post-Baseline value [week 4]) minus log (Baseline value).
Time Frame: Baseline (Week 0, Visit 2) and Week 4
Population: Full Analysis Set (FAS) Population was defined as all randomized participants who received at least one dose of study medication during treatment period and who had at least one evaluable assessment of Lp-PLA2 activity after randomization. Missing values during treatment period, except for Baseline were imputed by last observed response (LOCF).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Log(millimole per milliliter per minute)
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg
Number analyzed (Participants) | 25 | 28 | 28 | 26
Log(millimole per milliliter per minute) | 0.961 (8.5) | 0.494 (24.6) | 0.404 (21.5) | 0.313 (24.7)
Statistical Analysis 1: Comparison: Placebo vs SB-480848 40 mg; Test type: Superiority; p < .001, ANCOVA; Ratio = 0.514, 95% CI 2-sided [0.449 to 0.590] — The point estimate was calculated as adjusted geometric mean ratio of placebo and SB-480848 40 mg. Dunnett adjustment was used for comparison of each dose group to placebo
Statistical Analysis 2: Comparison: Placebo vs SB-480848 80 mg; Test type: Superiority; p < .001, ANCOVA; Ratio = 0.421, 95% CI 2-sided [0.367 to 0.483] — The point estimate was calculated as adjusted geometric mean ratio of placebo and SB-480848 80 mg. Dunnett adjustment was used for comparison of each dose group to placebo
Statistical Analysis 3: Comparison: Placebo vs SB-480848 160 mg; Test type: Superiority; p < .001, ANCOVA; Ratio = 0.326, 95% CI 2-sided [0.284 to 0.375] — The point estimate was calculated as adjusted geometric mean ratio of placebo and SB-480848 160 mg. Dunnett adjustment was used for comparison of each dose group to placebo

2. Secondary Outcome: Percent Inhibition of Lp-PLA2 Activity in Plasma Over Time
Description: Blood sample for Lp-PLA2 activity was collected before administration of study medication on the sampling day. Participants were instructed to visit without meal and study medication in the morning. The study medication was administered with food following test. Baseline value was defined as the assessment done on Week 0 (Visit 2). Percentage inhibition of Lp-PLA2 activity relative to a Baseline value was calculated as: 100 multiplied by (post-Baseline values (Week 1, 2, 4 and Follow-up-Baseline value) divided by [Baseline value]).
Time Frame: Baseline (Week 0, Visit 2) up to Follow-up (up to Week 7)
Population: FAS Population with LOCF analysis.
Measure: Mean (Standard Deviation); unit: Percent inhibiton of Lp-PLA2 activity
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg
Number analyzed (Participants) | 25 | 28 | 28 | 26
Percent inhibiton of Lp-PLA2 activity
  Week 1 | -4.06 (7.025) | -48.25 (15.929) | -55.83 (11.031) | -66.03 (7.656)
  Week 2 | -1.96 (8.147) | -49.05 (11.094) | -58.95 (8.258) | -67.52 (9.402)
  Week 4 | -3.59 (7.822) | -49.05 (13.472) | -58.67 (9.438) | -67.73 (8.310)
  Week 7 (Follow-up) | -3.16 (9.018) | -7.65 (11.408) | -9.40 (8.667) | -13.36 (10.244)

3. Secondary Outcome: Change From Baseline in Lp-PLA2 Activity at Week 1, 2 and Follow-up
Description: Blood sample for Lp-PLA2 activity was collected before administration of study medication on the sampling day. Participants were instructed to visit without meal and study medication in the morning. The study medication was administered with food following test. Baseline value was defined as the assessment done on Week 0 (Visit 2). Change from Baseline was calculated as the post-Baseline (Week 1, Week 2 and Follow-up) assessment values minus the Baseline assessment value. If either value was missing, then the change from Baseline was set to be missing. The log was used for transformation in Lp-PLA2 activity. In case of zero values, an offset of 0.0001 was added to the zero values to ensure that the log transformation was successfully applied. The log transformation was conducted on the original value and then taken change from Baseline on that log original value, calculated as log (post-Baseline [Week 1, Week 2 and Follow-up] values) minus log (Baseline value).
Time Frame: Baseline (Week 0, Visit 2), Week 1, Week 2 and Follow-up ( Week 7)
Population: FAS Population with LOCF analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Log(millimole per milliliter per minute)
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg
Number analyzed (Participants) | 25 | 28 | 28 | 26
Log(millimole per milliliter per minute)
  Week 1 | 0.957 (7.4) | 0.495 (30.9) | 0.430 (24.1) | 0.332 (22.5)
  Week 2 | 0.977 (8.4) | 0.499 (20.9) | 0.403 (19.0) | 0.313 (28.3)
  Week 7 (Follow-up) | 0.964 (9.6) | 0.917 (11.6) | 0.902 (9.8) | 0.860 (12.1)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded up to Follow-up (up to Week 7).
Description: Safety Population comprised of all participants who received at least one dose of the study medication during the treatment period.
Arm/Group | Placebo | SB-480848 40 mg | SB-480848 80 mg | SB-480848 160 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28 | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/28 | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 8/25 | 12/28 | 13/28 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | SB-480848 40 mg (N=28) | SB-480848 80 mg (N=28) | SB-480848 160 mg (N=26)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | SB-480848 40 mg (N=28) | SB-480848 80 mg (N=28) | SB-480848 160 mg (N=26)
Abnormal faeces (Gastrointestinal disorders) | 0 | 5 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 2 | 5 | 4
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.